CLINICAL TRIAL: NCT00911963
Title: A Phase l b/II a, Multicenter, Randomized, Double-Blinded, and Placebo-Controlled Study of the Antiviral Activity, Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of VCH-222 in Subjects With Chronic Hepatitis C-Infection
Brief Title: Pharmacokinetics of Multiple Ascending Doses of VCH-222 in Subjects With Chronic Hepatitis C Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: ViroChem Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCH-222-102
Record Dates: First submitted 2009-05-29; First posted 2009-06-03 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-02

CONDITIONS: Hepatitis C
Keywords: VX-222
MeSH Terms: conditions — Hepatitis C | interventions — lomibuvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Experimental): This will be a 4 dose escalation study comparing VCH-222 to placebo treatment.
  Interventions: Drug: VCH-222 or matching placebo
- Part B (Experimental): VCH-222 + peginterferon alfa-2a + ribavirin (12 weeks) followed by peginterferon alfa-2a + ribavirin for 36 weeks
  Interventions: Drug: VCH-222 or matching placebo; Biological: peginterferon alfa-2a; Drug: ribavirin

INTERVENTIONS:
Drug: VCH-222 or matching placebo — capsule, oral, 4 doses once daily or twice daily, 3 days
  Other Names: VCH-222 is also known as VX-222
  Arms: Part A
Drug: VCH-222 or matching placebo — capsule, oral, 400 mg twice daily or 750 mg twice daily, 12 weeks
  Other Names: VCH-222 is also known as VX-222
  Arms: Part B
Biological: peginterferon alfa-2a — subcutaneous injection, 180 μg, once weekly, 48 weeks
  Arms: Part B
Drug: ribavirin — tablet, oral, 1000-1200 mg daily based on body weight, 48 weeks
  Arms: Part B

SUMMARY:
The purpose of this study is to assess antiviral activity when administered alone for 3 days or in combination with peginterferon and ribavirin for 12 weeks. This study will also evaluate the safety and tolerability of treatment with VCH-222 when given alone or in combination with peginterferon and ribavirin.

The study will also evaluate the pharmacokinetic profile of VCH-222 in HCV infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects, 18-65 years of age (females non-child bearing potential in Part B)
* Have laboratory evidence of HCV infection for 6 months, defined by (1) presence of anti-HCV antibody (Genotype 1a and 1b infection), or (2)documented HCV RNA presence by a sensitive and specific assay and (3 histologic evidence of CHC (Fibrosis on a standardized histological grading system)
* Plasma HCV RNA of 100,000 IU/ml
* HIV 1 and HIV2 ab seronegative
* Body Mass Index (BMI) ≤ 35 kg/m2 BMI
* Treatment Naive subjects

Exclusion Criteria:

* Contraindications to peginterferon or ribavirin therapy
* Have evidence of liver cirrhosis, decompensated liver disease, and Child-Pugh score > 5
* Have hemoglobinopathies, unstable cardiac disease, history of organ transplant, active malignant disease or uncontrolled Type I or II diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To assess the antiviral activity of VCH-222, in subjects with genotype 1 hepatitis C virus (HCV) infection after once (QD) or twice (b.i.d.) daily dosing for 3 days (Part A) | Daily for the first 3 days and at each study visit
To assess the antiviral activity of VCH-222, in subjects with genotype 1 HCV infection after b.i.d. daily dosing for 12 weeks in combination with Peg-interferon-alfa-2a and ribavirin (Part B) | Week 4 and Week 12
Assess the safety and tolerability of VCH-222 when administered in combination with Peg-IFN-alfa-2a/RBV for 12 weeks (Part B) | Study visits throughout part B

SECONDARY OUTCOMES:
To assess the safety and tolerability of VCH-222 when administered for 3 days in monotherapy (Part A) | Study visits throughout Part A
To evaluate the pharmacokinetic (PK) profile of VCH-222 in HCV infected subjects (Part B) | Time points through Part B

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (10):
- United States (4):
  - Gastrointestinal Specialists of Georgia PC, Marietta, Georgia
  - Henry Ford Health Sytem, Detroit, Michigan
  - The liver institute at Methodist hospital, Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas
- Argentina (2):
  - ACLIRES Argentina SRL, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
- Canada (3):
  - Downtown ID Clinic/University of British Columbia, Vancouver, British Columbia
  - John Buhler Research Centre, Winnipeg, Manitoba
  - Ottawa Hospital, Ottawa, Ontario
- Fundacion de Investigation de Diego, Santurce, Puerto Rico

REFERENCES:
- [Derived] Jiang M, Zhang EZ, Ardzinski A, Tigges A, Davis A, Sullivan JC, Nelson M, Spanks J, Dorrian J, Nicolas O, Bartels DJ, Rao BG, Rijnbrand R, Kieffer TL. Genotypic and phenotypic analyses of hepatitis C virus variants observed in clinical studies of VX-222, a nonnucleoside NS5B polymerase inhibitor. Antimicrob Agents Chemother. 2014 Sep;58(9):5456-65. doi: 10.1128/AAC.03052-14. Epub 2014 Jun 30. PMID 24982088